CLINICAL TRIAL: NCT01304342
Title: The Effect of Intranasal Fentanyl Versus Remifentanil Infusion on Propofol Requirements During Elective Therapeutic ERCP, as Well on the Recovery, Pain, and Early Cognitive Function: A Randomized Control Trial
Brief Title: Sedation in Endoscopic Retrograde Cholangiopancreatography (ERCP) With or Without Opioids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Argyro Fassoulaki, MD, PhD, DEAA, University of Athens
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M-17, M-18/21-12-2010
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2012-03

CONDITIONS: Chronic Pain
Keywords: Propofol; remifentanil; fentanyl; ERCP; Quality of sedation; recovery; satisfaction; respiratory depression
MeSH Terms: conditions — Chronic Pain; Personal Satisfaction; Respiratory Insufficiency | interventions — Remifentanil; Fentanyl; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Remifentanil (Active Comparator): Remifentanil 1 microgram/kg/h along with propofol infusion
  Interventions: Drug: Remifentanil
- Fentanyl (Active Comparator): Fentanyl 200 micrograms intranasally
  Interventions: Drug: Fentanyl
- Normal saline (Placebo Comparator): Normal saline intravenously and intranasally
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Remifentanil — 1 microgram/kg/h, continuous infusion, 5 min before and during the ERCP
  Other Names: Ultiva
  Arms: Remifentanil
Drug: Fentanyl — Intranasal fentanyl 200 micrograms 5 min before the ERCP
  Arms: Fentanyl
Drug: Normal saline — Normal saline intravenously and intranasally
  Arms: Normal saline

SUMMARY:
Addition of fentanyl or remifentanil to the propofol produced sedation for scheduled ERCP will decrease the propofol requirements for predetermined sedation levels (as shown by Bispectral Index Monitor (BIS) monitor), will be associated with faster recovery monitored by Ramsay's and Observer's Assessment of Alertness/Sedation (OAAS) scores and BIS, less postoperative pain (assessed by Visual Analogue Scale=VAS) and less early cognitive impairment after sedation (as assessed by the MiniMental test).

DETAILED DESCRIPTION:
Patients After obtaining approval from the Institutional Review Board (IRB) adult patients ASA I-III aged between 45 and 75 yrs scheduled for elective therapeutic ERCP are enrolled in the study. All patients are informed and asked to give written informed consent. Those with chronic pain, consuming opioids or other analgesics, sedatives, hypnotics, allergic to the drugs to be used in the study protocol, or patients who refuse to give written informed consent are excluded from the study.

Randomization and blindness Randomization was done by a Research Randomizer program, using 60 sets of numbers and 3 numbers per set for a total of 180 patients, keeping each number in a set to remain unique and without sorting the numbers that are generated. (http://www.randomizer.org/). The remifentanil or placebo solutions as well as the nasal fentanyl or placebo spray are prepared and administered by an independent investigator who is aware of the group randomization and indicated interventions.

Group 1: Receive remifentanil i.v infusion 1 ml/10 kg/h (10 μg/ml) starting 5 minutes before propofol administration and continued throughout the procedure. At the same time intranasal normal saline is given. A bolus dose of propofol 1 mg/kg is followed by propofol infusion and the infusion is titrated to obtain BIS values around 40-70.

Group 2: Receive normal saline i.v. infusion in volume equal to the volume of remifentanil as if he/she were assigned to Group 1, intranasal fentanyl 200 μg, and propofol as in group 1.

Group 3: Receive i.v. normal saline infusion in volume equal to the volume of remifentanil as if he/she were assigned to Group 1, intranasal normal saline, and propofol as in groups 1 and 2.

Anesthetic technique Before opioid/placebo/anesthetic administration all patients receive for 3-5 min 100% oxygen via a face mask from a wall oxygen source by means of a Mapleson C breathing system. Two venous catheters are inserted in peripheral veins and connected via extension tubes to two separate infusion pumps for remifentanil or placebo and for propofol infusion.

Basic monitoring includes pulse oximetry, non-invasive blood pressure (measured in the beginning and at the end of the procedure), heart rate, respiratory rate and ECG. Additional monitoring includes BIS, (BIS VIEW ™ Monitoring System, Aspect Medical Systems, Inc. One Upland Road Norwood, MA 02062 USA). All patients are preoxygenated with 100% oxygen via a face mask before anesthetic administration. During the procedure oxygen (9 l/min) is administered via a nasal catheter. Sedation/anesthesia is maintained with propofol bolus 1 mg/kg to begin with, plus infusion (5-9 mg/kg/h) by means of an electric pump to obtain BIS values around 40-70.

Intraoperative variables to be recorded Baseline values (before starting opioid/placebo) and every 3 min thereafter throughout the procedure BIS, SpO2, HR, RR, and Movement of the patient (Yes/No) are recorded and the propofol infusion is increased accordingly. Systolic and diastolic blood pressure is recorded in the beginning and at the end of the procedure (not to disturb the patient and change the level of consciousness, except for complications during the procedure like bleeding, apnea etc). Also events of desaturation (SpO2 below 90), episodes of apnea (apnea for > than 30s), and other adverse events are recorded. Systolic and diastolic blood pressure is recorded in the beginning and at the end of the procedure (not to disturb the patient and change the level of consciousness, except for complications during the procedure, like bleeding, apnea etc).

At the end of the procedure the total doses of propofol and remifentanil (or the volume of placebo) are recorded.

ELIGIBILITY:
Inclusion Criteria:

* patients both sexes
* ASA I-III
* aged between 45 and 75 years old
* scheduled for interventional ERCP

Exclusion Criteria:

* patients receiving opioids or other analgesics, sedatives, hypnotics
* allergic to drugs used in the study protocol
* alcoholism
* refuse to sign the informed consent and chronic pain

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2011-02; Primary Completion 2013-01 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Propofol requirements | 30 min, 60 min and if not full recovery 120 min

SECONDARY OUTCOMES:
Speed of recovery | 30, 60 and 120 min
postoperative pain | 30, 60, and 120 minutes
early cognitive function | 30, 60, and 120 minutes
patient satisfaction | 30, 60, and 120 minutes
endoscopist satisfaction | 30, 60, and 120 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Aretaieio Hospital, Athens, Greece

REFERENCES:
- [Derived] Fassoulaki A, Iatrelli I, Vezakis A, Polydorou A. Deep sedation for endoscopic cholangiopancreatography with or without pre or intraprocedural opioids: A double-blind randomised controlled trial. Eur J Anaesthesiol. 2015 Sep;32(9):602-8. doi: 10.1097/EJA.0000000000000187. PMID 25405276